CLINICAL TRIAL: NCT06226220
Title: Trial Time for Percutaneous Nerve Evaluation in Patients Undergoing Sacral Neuromodulation for Urgency Urinary Incontinence or Urgency-frequency: a Randomized Control Trial
Brief Title: Percutaneous Nerve Evaluation Trial Time
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Allegheny Health Network (Other); University of California, Irvine (Other); Atrium Health Wake Forest Baptist (Other); University of Texas (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0942
Record Dates: First submitted 2023-12-12; First posted 2024-01-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Urge Incontinence; Urgency-frequency Syndrome; Overactive Bladder
Keywords: urinary urgency; urinary incontinence; urinary frequency; overactive bladder; sacral neuromodulation; percutaneous nerve evaluation
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, non-inferiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 3-day trial (Experimental): Patients randomized to the 3-day trial arm will undergo a 3-day PNE trial phase for sacral neuromodulation. Participants will have the PNE placed in the office and return on day 3 for PNE removal.
  Interventions: Procedure: Sacral neuromodulation
- 7-day trial (Active Comparator): Patients randomized to the73-day trial arm will undergo a 7-day PNE trial time for sacral neuromodulation. Participants will have the PNE placed in the office and return on day 7 for PNE removal.
  Interventions: Procedure: Sacral neuromodulation

INTERVENTIONS:
Procedure: Sacral neuromodulation — Sacral neuromodulation (SNM) is a minimally invasive procedure that provides low-amplitude electrical stimulation to the S3 nerve root to improve micturition and defecation. Patients who elect to proceed with SNM undergo a trial phase to determine therapeutic response prior to placement of a permanent implantable pulse generator (IPG). A trial phase can be performed in two ways: a percutaneous nerve evaluation (PNE) or staged implantation. PNE involves the placement of a temporary wire connected to an electrode using external stimulation. It is performed in the office using local anesthesia. If the patient displays adequate improvement in symptoms (defined as >50% improvement of symptoms from baseline), a permanent lead and subcutaneous IPG are implanted in the operating room.
  Other Names: Percutaneous nerve evaluation

SUMMARY:
Sacral neuromodulation (SNM) was approved by the Food and Drug Administration (FDA) for the treatment of urgency incontinence (UUI) in 1998. One of two trial phase techniques are utilized prior to placement of the implantable pulse generator (IPG) to predict a patient's success with the device: a percutaneous nerve evaluation (PNE) or a stage implantation. Patients who experience a > 50% improvement in UUI symptoms progress to permanent implantation. PNE offers significant advantages compared to a staged implantation including a single anesthetic and operating room trip. Historically, full implantation rates are only 40-50% following PNE versus 70-90% in women who undergo a staged approach. The lower rate of progression to full implantation after PNE may be attributed to lead migration. Newer data suggest up to 90% of PNE trials lead to full implantation. The investigators hypothesize that shortening PNE trial time to 3 days from 7 days will not result in a lower proportion of PNE trials leading to SNM implantation and may offer less time for lead migration. The investigators aim to perform a multi-center, randomized trial to determine if a 3-day PNE trial is not inferior to a 7-day PNE trial with respect to rates of progression to SNM implantation.

DETAILED DESCRIPTION:
Sacral neuromodulation (SNM) is a minimally invasive procedure that provides low-amplitude electrical stimulation to the S3 nerve root to improve micturition and defecation. It is FDA-approved for the treatment of urgency urinary incontinence (UUI) refractory to behavioral modifications and/or oral medication. The efficacy of SNM for the treatment of UUI is well studied and currently, there are two manufacturers of SNM devices within the United States: Medtronic and Axonics. Both offer rechargeable and non-rechargeable devices.

Patients who elect to proceed with SNM undergo a trial phase to determine therapeutic response prior to placement of a permanent implantable pulse generator (IPG). A trial phase can be performed in two ways: a percutaneous nerve evaluation (PNE) or staged implantation. PNE involves the placement of a temporary wire connected to an electrode using external stimulation. It is performed in the office using local anesthesia. If the patient displays adequate improvement in symptoms (defined as >50% improvement of symptoms from baseline), a permanent lead and subcutaneous IPG are implanted in the operating room. The staged approach involves two separate procedures performed in the operating room: stage I and stage II. Stage I is the clinical trial of the permanent lead with electrodes using external stimulation. Following adequate response, stage II is performed and involves the IPG placement.

PNE offers significant advantages compared to a staged implantation. A PNE is performed in the office under local anesthesia mitigating the anesthetic risk and number of operating room visits. PNE is also suspected to be cost-effective given it is performed in the office with minimal medical equipment; however, this has not been well studied. Full implantation rates are 40-50% following PNE versus 70-90% in women who undergo a staged approach. The lower rate of progression to full implantation with PNE can be attributed to several factors including lead migration. The monopolar PNE lead does not have a self-retaining component like the quadripolar tined lead used during a stage approach. Newer registry data suggest up to 90% of PNE trials lead to full implantation. Authors hypothesize the improved full implantation rates in the newer studies may be secondary to shorter trial times and improved anatomic knowledge.

The trial phase is the most valuable tool to predict therapeutic success of SNM for women with UUI. Several large, multicenter trials support that PNE and staged trial can predict patients who are likely to respond to SNM therapy and experience long term benefits. Literature is limited regarding recommended length of time for the trial phase. The International Continence Society best practice statement for use of SNM currently recommends 7-day trial for women with UUI. However, one study reported high sensitivity and specificity of PNE with a trial time of 3-5 days. This cross-sectional study was limited to a single institution and included patients with nonobstructive urinary retention.

Given the risk of lead migration with PNE, the investigators hypothesize that shortening the trial phase to 3 days will not decrease the proportion of patients who progress onto full SNM implantation. The investigators believe that shortening the window to capture therapeutic response will have several important patient benefits and reduce the chance of lead migration without adversely impacting outcomes. Therefore, the investigators aim to perform a multi-center, randomized trial to determine if a 3-day PNE trial is not inferior to a 7-day PNE trial with respect to rates of progression to full SNM implantation.

The investigators plan to perform a multi-center, randomized, non-inferiority trial of patients receiving SNM for UUI or urgency-frequency syndrome (UF) who elect to undergo a PNE. Informed consent will be obtained for participants who meet eligibility criteria. Participants will be computer randomized in a 1:1 fashion to either a 3 or 7-day PNE trial on the day of PNE (to minimize bias and drop out). Permuted blocks will be utilized with a fixed block size stratified by age (<65 versus >65 years old) and study site. Decision to stratify by age is based on the association between advancing age and decreased SNM response. Patients must have at least 5 episodes of UUI or at least 8 voids per day for 2 days on a 3-day bladder diary to be included. Demographic and symptom data will be collected at participants baseline visit including a 3-day bladder diary and validated patient reported outcome measures for urinary symptoms and quality of life (Urinary Distress Inventory, Lower Urinary Tract Dysfunction Research Network Symptom Index-10, Incontinence Impact Questionnaire). At the PNE visit and PNE removal, clinical information will be recorded, and patient reported outcome measures will be repeated (including Patient Global Impression of Improvement). Patients who have an adequate response to PNE placement (>50% improvement in UUI/UF symptoms determined by 3-day bladder diary) will progress to full SNM implantation.

Assuming a significance level of 5% and 80% rate of progression to full implantation in each arm with a noninferiority margin of 15 percentage points, the investigators calculate that 88 women would need to enroll in each study arm to have 80% power for determining whether the results in the 3-day PNE trial arm are noninferior to those in the 7-day trial arm. The investigators propose a 15% noninferiority margin on the basis of clinical judgement that this is a reasonable tradeoff between a decrease in progression to full or stage implantation and the possibility of shortening the PNE trial period. Assuming a 10% dropout rate, a total sample of 193 women will be required. Non-inferiority will be declared if the upper bound of the 95% confidence interval for the rate of progression to full implantation between groups is less than 15%. To minimize bias toward noninferiority, only women treated per protocol will be considered in the primary outcome analysis.

De-identified data will be collected at each site in a REDCap database then transferred to an SPSS database (IBM SPSS Statistics for Macintosh, Version 22.0. Armonk, NY: IBM Corp) for statistical analysis. Secondary outcomes will be assessed using intent to treat analyses.

Comparative statistics for patient demographics and clinical outcomes will be performed between the two cohorts utilizing chi-square, t-test, and Wilcoxon test as appropriate for continuous and categorical variables. Logistic regression models will be used to evaluate the association between factors and rate of full SNM implantation following PNE. Multivariate logistic regression to control for potential cofounding variables.

The investigators estimate being able to recruit 3 women undergoing PNE each month during the study period from the investigator's site or 36 participants in 1-year. Given the standard of care is a 7-day PNE, the investigators anticipate patients will be eager for the option to be randomized to a less onerous test period. In addition, the only patient burden (beyond standard of care) is completion of a series of validated questionnaires, which the investigators estimate will take 15 minutes at both time points. There are currently two SNM device manufacturers (Medtronic and Axonics) as well as a national-reported increased in SNM implantation procedures over the past decade.15 While there are no comparative date between these devices, the investigators think both can be included in this trial to increase generalizability.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women >/=18 years old undergoing sacral neuromodulation (SNM) treatment for urgency urinary incontinence (UUI) or urgency-frequency (UF) who have elected to undergo testing phase with a PNE
* >/=5 UUI episodes on a 3-day bladder diary with urge incontinence representing >/=50% of total incontinence episodes recorded or >/=8 per day for 2 days on a 3-day bladder diary
* Willing and able to complete all study related items and interviews
* Grossly neurologically normal exam

Exclusion Criteria:

* SNM indication of non-obstructive urinary retention or isolated fecal incontinence
* Severe or poorly controlled diabetes (defined as HgbA1c >/=8.0) or diabetes with peripheral nerve involvement
* Neurological diseases such as multiple sclerosis, clinically significant peripheral neuropathy, or complete spinal cord injury
* Surgically altered detrusor muscle (i.e. Augmentation cystoplasty)
* Current or prior bladder malignancy
* Prior pelvic irradiation
* Post void residual (PVR) >/= 150 mL within 6 months prior to enrollment
* Active urinary tract infection
* Primary stress urinary incontinence or mixed urinary incontinence with stress predominance
* >/= Stage III pelvic organ or vaginal vault prolapse and/or current pessary use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of progression onto full sacral neuomodulation (SNM) implant | 3 or 7 days depending on treatment arm
  Participants with an adequate therapeutic response during percutaneous nerve evaluation (PNE) trial (>/=50% improvement in urgency urinary incontinence (UUI)/ urgency-frequency (UF) symptoms) will progress onto full SNM implantation

SECONDARY OUTCOMES:
Patient satisfaction | 3 or 7 days depending on treatment arm
  Participants will complete validated patient reported outcome measures at baseline and at PNE lead pull
Rate of adverse events | 3 or 7 days depending on treatment arm
  Adverse events during trial phase will be recorded
Quality of life scores | 3 or 7 days depending on treatment arm
  Participants will complete validated patient reported outcome measures at baseline and at PNE lead pull

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kenton, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel S, Noblett K, Mangel J, Griebling TL, Sutherland SE, Bird ET, Comiter C, Culkin D, Bennett J, Zylstra S, Berg KC, Kan F, Irwin CP. Results of a prospective, randomized, multicenter study evaluating sacral neuromodulation with InterStim therapy compared to standard medical therapy at 6-months in subjects with mild symptoms of overactive bladder. Neurourol Urodyn. 2015 Mar;34(3):224-30. doi: 10.1002/nau.22544. Epub 2014 Jan 10. PMID 24415559
- [Background] Amundsen CL, Komesu YM, Chermansky C, Gregory WT, Myers DL, Honeycutt EF, Vasavada SP, Nguyen JN, Wilson TS, Harvie HS, Wallace D; Pelvic Floor Disorders Network. Two-Year Outcomes of Sacral Neuromodulation Versus OnabotulinumtoxinA for Refractory Urgency Urinary Incontinence: A Randomized Trial. Eur Urol. 2018 Jul;74(1):66-73. doi: 10.1016/j.eururo.2018.02.011. Epub 2018 Feb 24. PMID 29482936
- [Background] Bannowsky A, Wefer B, Braun PM, Junemann KP. Urodynamic changes and response rates in patients treated with permanent electrodes compared to conventional wire electrodes in the peripheral nerve evaluation test. World J Urol. 2008 Dec;26(6):623-6. doi: 10.1007/s00345-008-0307-7. Epub 2008 Jul 16. PMID 18629503
- [Background] Hijaz A, Vasavada SP, Daneshgari F, Frinjari H, Goldman H, Rackley R. Complications and troubleshooting of two-stage sacral neuromodulation therapy: a single-institution experience. Urology. 2006 Sep;68(3):533-7. doi: 10.1016/j.urology.2006.03.020. Epub 2006 Sep 18. PMID 16979724
- [Background] Blandon RE, Gebhart JB, Lightner DJ, Klingele CJ. Re-operation rates after permanent sacral nerve stimulation for refractory voiding dysfunction in women. BJU Int. 2008 May;101(9):1119-23. doi: 10.1111/j.1464-410X.2007.07426.x. Epub 2008 Jan 10. PMID 18190624
- [Background] Borawski KM, Foster RT, Webster GD, Amundsen CL. Predicting implantation with a neuromodulator using two different test stimulation techniques: A prospective randomized study in urge incontinent women. Neurourol Urodyn. 2007;26(1):14-8. doi: 10.1002/nau.20332. PMID 17123297
- [Background] Spinelli M, Weil E, Ostardo E, Del Popolo G, Ruiz-Cerda JL, Kiss G, Heesakkers J. New tined lead electrode in sacral neuromodulation: experience from a multicentre European study. World J Urol. 2005 Jul;23(3):225-9. doi: 10.1007/s00345-005-0502-8. Epub 2005 Jun 30. PMID 15988594
- [Background] Siegel SW, Catanzaro F, Dijkema HE, Elhilali MM, Fowler CJ, Gajewski JB, Hassouna MM, Janknegt RA, Jonas U, van Kerrebroeck PE, Lycklama a Nijeholt AA, Oleson KA, Schmidt RA. Long-term results of a multicenter study on sacral nerve stimulation for treatment of urinary urge incontinence, urgency-frequency, and retention. Urology. 2000 Dec 4;56(6 Suppl 1):87-91. doi: 10.1016/s0090-4295(00)00597-5. PMID 11114569
- [Background] Al-zahrani AA, Elzayat EA, Gajewski JB. Long-term outcome and surgical interventions after sacral neuromodulation implant for lower urinary tract symptoms: 14-year experience at 1 center. J Urol. 2011 Mar;185(3):981-6. doi: 10.1016/j.juro.2010.10.054. Epub 2011 Jan 19. PMID 21247597
- [Background] Goldman HB, Lloyd JC, Noblett KL, Carey MP, Castano Botero JC, Gajewski JB, Lehur PA, Hassouna MM, Matzel KE, Paquette IM, de Wachter S, Ehlert MJ, Chartier-Kastler E, Siegel SW. International Continence Society best practice statement for use of sacral neuromodulation. Neurourol Urodyn. 2018 Jun;37(5):1823-1848. doi: 10.1002/nau.23515. Epub 2018 Apr 11. PMID 29641846
- [Background] Banakhar M, Hassouna M. Percutaneous Nerve Evaluation Test Versus Staged Test Trials for Sacral Neuromodulation: Sensitivity, Specificity, and Predictive Values of Each Technique. Int Neurourol J. 2016 Sep;20(3):250-254. doi: 10.5213/inj.1630498.249. Epub 2016 Sep 23. PMID 27706006
- [Background] Amundsen CL, Romero AA, Jamison MG, Webster GD. Sacral neuromodulation for intractable urge incontinence: are there factors associated with cure? Urology. 2005 Oct;66(4):746-50. doi: 10.1016/j.urology.2005.04.031. PMID 16230129
- [Background] White WM, Mobley JD 3rd, Doggweiler R, Dobmeyer-Dittrich C, Klein FA. Sacral nerve stimulation for refractory overactive bladder in the elderly population. J Urol. 2009 Oct;182(4):1449-52. doi: 10.1016/j.juro.2009.06.049. Epub 2009 Aug 15. PMID 19683295
- [Background] Elterman DS, Chughtai B, Vertosick E, Thomas D, Eastham J, Sandhu J. Trends and Clinical Practice Patterns of Sacral Neuromodulation for Overactive Bladder. Female Pelvic Med Reconstr Surg. 2018 Jul/Aug;24(4):264-266. doi: 10.1097/SPV.0000000000000449. PMID 28658001